CLINICAL TRIAL: NCT01515163
Title: Exercise and Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, PhD, Assistant Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lupus and exercise
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise (Experimental): 3-month exercise training program
  Interventions: Behavioral: Exercise training
- Control (No Intervention): Control group
- Healthy control (Experimental)
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Aerobic exercise training, two times a week
  Arms: Exercise; Healthy control

SUMMARY:
The investigators hypothesize that a three-month aerobic exercise training program will positively affect the lipid profile, insulin sensitivity , cytokine profile, the cardiovascular parameters and muscle strength in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 and 40 years
* SLEDAI ≤ 4

Exclusion Criteria:

* Cardiovascular dysfunction
* Rhythm and conduction disorders
* Musculoskeletal disturbances
* Kidney and pulmonary involvements
* Peripheral neuropathy
* Use of tobacco
* Treatment with lipid-lowering or hypoglycemic drugs
* Fibromyalgia
* Use of chronotropic or antihypertensive drugs
* Physically active subjects

Ages: 7 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2010-05; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Lipid profile - Plasma levels of total cholesterol (mg/dl), VLDL-chol (mg/dl) HDL-chol (mg/dl), LDL-chol (mg/dl), triglycerides (mg/dl), Apolipoprotein AI and AII (mg/dl) and Apolipoprotein B (mg/dl) | 3 months
Insulin sensitivity as measured by the Hyperinsulinemic-Euglycemic Clamp | 3 months
Cytokine response - Plasma levels of TNF-α (pg/ml), IL-6 (pg/ml), IFN-type I (pg/ml), IL-10 (pg/ml)and IL-1ra (pg/ml) | 3 months

SECONDARY OUTCOMES:
Cardiovascular parameters | 3 months
  Aerobic capacity, chronotropic function
Muscle Strength | 3 months
  Upper and Lower-body muscle strength will be assessed by a 1-RM (repetition maximum) protocol

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Benatti FB, Miyake CNH, Dantas WS, Zambelli VO, Shinjo SK, Pereira RMR, Silva MER, Sa-Pinto AL, Borba E, Bonfa E, Gualano B. Exercise Increases Insulin Sensitivity and Skeletal Muscle AMPK Expression in Systemic Lupus Erythematosus: A Randomized Controlled Trial. Front Immunol. 2018 Apr 27;9:906. doi: 10.3389/fimmu.2018.00906. eCollection 2018. PMID 29755474
- [Derived] Benatti FB, Miossi R, Passareli M, Nakandakare ER, Perandini L, Lima FR, Roschel H, Borba E, Bonfa E, Gualano B, de Sa Pinto AL. The effects of exercise on lipid profile in systemic lupus erythematosus and healthy individuals: a randomized trial. Rheumatol Int. 2015 Jan;35(1):61-9. doi: 10.1007/s00296-014-3081-4. Epub 2014 Jun 28. PMID 24972700
- [Derived] Prado DM, Benatti FB, de Sa-Pinto AL, Hayashi AP, Gualano B, Pereira RM, Sallum AM, Bonfa E, Silva CA, Roschel H. Exercise training in childhood-onset systemic lupus erythematosus: a controlled randomized trial. Arthritis Res Ther. 2013 Mar 26;15(2):R46. doi: 10.1186/ar4205. PMID 23531226